CLINICAL TRIAL: NCT07119489
Title: A Novel Dialectical Behavior Therapy Brief Group Intervention for Cigarette Smoking by Patients With Cancer: An Open Clinical Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Atrium Health Wake Forest Baptist (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00131890; ONC-CCS-2408 (Other: Atrium Health Wake Forest Baptist Comprehensive Cancer Center)
Record Dates: First submitted 2025-07-28; First posted 2025-08-13 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-07

CONDITIONS: Smoking Behavior
Keywords: Dialectical Behavior Therapy; Cancer; Smoking
MeSH Terms: conditions — Smoking; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with cancer who smoke (Experimental): Participants who smoke and are undergoing treatment with a curative intent for cancer or are in remission from cancer
  Interventions: Behavioral: Dialectical Behavior Therapy -Skill Training brief intervention

INTERVENTIONS:
Behavioral: Dialectical Behavior Therapy -Skill Training brief intervention — A behavioral counseling approach for enhancing skills in emotion regulation, distress tolerance, and mindfulness

SUMMARY:
The purpose of this research study is to learn more about how Dialectical Behavior Therapy - Skills Training can help patients with cancer who smoke cigarettes cut down on or stop their smoking.

DETAILED DESCRIPTION:
This is a study that aims to evaluate recruitment rates, feasibility, acceptability, and fidelity of Dialectical Behavior Therapy - Skills Training (DBT-ST) brief intervention.

Study population will include participants who smoke and are undergoing treatment with curative intent for their cancer or are in remission.

The study will include eight 60 minute sessions of DBT-ST and measurements of psychological states and smoking habits by interventionists. At follow-up participants will complete a survey on their intervention experience and ongoing use of DBT-ST. Interventionists will also complete a survey following each session to record time and materials use for future cost-effectiveness analysis.

At follow-up, participants and interventionists will engage in a one-hour qualitative interview with a study team member.

ELIGIBILITY:
Inclusion Criteria:

1. Smoke ≥1 cigarettes every day in the past 30 days per participant report.
2. Smoked at least 100 cigarettes (5 packs) in lifetime.
3. Confirmation of cancer and are in active treatment with curative intent or in remission per enrolling investigator or electronic medical record.
4. Age ≥ 18 years at the time of consent.
5. Ability to understand and willingness to sign an IRB-approved informed consent, in English, directly.
6. Able and willing to participate in video conference.

Exclusion Criteria:

1. Patients actively receiving external tobacco use counseling or using tobacco cessation medications.
2. Prior experience with more than five sessions of DBT-ST.
3. Life expectancy of six months or less.
4. Medical or psychiatric conditions limiting compliance with study requirements including suspected or reported cognitive impairment.
5. Self-reported use of any psychoactive substance [except marijuana and nicotine] within the last 30 days.
6. Have active and severe suicidal ideation at time of eligibility assessment or suicide attempt within the past month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Recruitment Rates | Measured from the date the first patient responds to advertisement or is referred to the study by providers until the date the last patient group begins the first session of the intervention, assessed up to 100 weeks.
  Ratio of patients enrolled in study to patients responding to advertisement or referred by providers, and ratio of patients enrolled to patients screened and potentially eligible for the study.
Feasibility of the DBT-ST brief intervention for cigarette smoking by patients with cancer | Measured from the date the first patient group begins the first session of the intervention until the date the last patient group completes the eighth session of the intervention, assessed up to 100 weeks.
  Rate of completion of the eight proposed sessions by participants
Acceptability of the DBT-ST brief intervention for cigarette smoking by patients with cancer | For each patient group, measured at weeks 1 through 8 of the intervention and at 1 month follow-up, assessed up to 100 weeks.
  Quantitative (Likert scale) questions to assess patient experience of intervention
Fidelity of the DBT-ST brief intervention for cigarette smoking by patients with cancer | Measured beginning 1 month after the date of week 8 of the final patient group participating in the intervention, assessed up to 6 months.
  Interventionist adherence to intervention manual will be assessed by having an independent reviewer select 50% of the audiotaped group sessions (the total depends on the number of groups) and complete a checklist of 25 intervention items (yes/no) to see whether the interventionist performed the item

SECONDARY OUTCOMES:
Cancer Patient Tobacco Use Questionnaire (C-TUQ) | Measured at baseline, week 5, week 8, and at 1 month follow-up, assessed up to 100 weeks.
  Changes in tobacco use, specifically number of days engaging in cigarette smoking (frequency) and number of cigarettes smoked per day (daily average) will be measured using the Cancer Patient Tobacco Use Questionnaire (C-TUQ) a 22-item self-report survey used to gather information about tobacco use by patients with cancer and cancer survivors.
Difficulties in Emotion Regulation Scale-36 (DERS-36) | Measured at baseline, week 5, week 8, and at 1 month follow-up, assessed up to 100 weeks.
  The Difficulties in Emotion Regulation Scale (DERS) is a 36-item self-report Likert scale used to assess emotional regulation presented as a total score and 6 sub-scores including nonacceptance of emotional responses, difficulty engaging in goal-directed behavior, impulse control difficulties, lack of emotional awareness, limited access to emotion regulation strategies, and lack of emotional clarity
Depression Anxiety Stress Scales-21 (DASS-21) | Measured at baseline, week 5, week 8, and at 1 month follow-up, assessed up to 100 weeks.
  The DASS-21 is a 21-item self-report instrument designed to measure the three related negative emotional states of depression, anxiety, and tension/stress.
Distress Tolerance Scale (DTS) | Measured at baseline, week 5, week 8, and at 1 month follow-up, assessed up to 100 weeks.
  Distress tolerance will be measured using the 15-item Distress Tolerance Scale (DTS). The DTS uses a 5-point Likert scale for participants to record responses to items (1 = 'Strongly Agree' to 5 = 'Strongly Disagree'). The total DTS score is calculated by adding the scores of all 15 items together after reverse-coding item 6 (score range 0-75)
Mindfulness Attention Awareness Scale (MAAS) | Measured at baseline, week 5, week 8, and at 1 month follow-up, assessed up to 100 weeks.
  Mindfulness will be measured using the Mindfulness Attention Awareness Scale (MAAS), a 15-item self-report instrument designed to assess a core characteristic of dispositional mindfulness, namely, open or receptive awareness of and attention to what is taking place in the present. The MAAS score is the mean of 15 Likert-scale items from 1-6 (score range 1-6)
Mental Adjustment to Cancer (MAC) Scale - Mini | Measured at baseline, week 5, week 8, and at 1 month follow-up, assessed up to 100 weeks.
  The MAC-Mini is a 29-item self-rating scale to assess psychological dimensions of in cancer patients of helplessness/hopelessness, anxious preoccupation, fatalism, avoidance, and fighting spirit in their adjustment to the diagnosis and treatment of cancer. Higher scores reflect lower levels of adjustment for all subscales except fighting spirit, with a higher score indicating higher adjustment
DBT Ways of Coping Checklist (DBT-WCCL) | Measured at baseline, week 5, week 8, and at 1 month follow-up, assessed up to 100 weeks.
  The DBT-WCCL is a 59-item self-report Likert scale, with one part assessing coping via DBT skills, the DBT Skills Subscale (DSS), and one part assessing coping via dysfunctional means, the Dysfunctional Coping Subscale (DCS).44 Skills use are measured on a scale from 0 (never used) to 3 (regularly used). Higher scores indicate more frequent use of DBT skills and functional coping behaviors.
Serious quit attempts | Measured at baseline, week 5, week 8, and at 1 month follow-up, assessed up to 100 weeks.
  The period of intentional abstinence from smoking typically lasting at least 24 hours, to be collected by self-report using a single item Serious Quit Attempt questionnaire

OTHER OUTCOMES:
Self-reported cost for interventionist and patient time and expenses | Measured at baseline, week 5, week 8, and at 1 month follow-up, assessed up to 100 weeks.
  Self-reported cost for interventionist and patient time and expenses will be collected using an interventionist questionnaire
Costs of nicotine replacement therapy | Measured at baseline, week 5, week 8, and at 1 month follow-up, assessed up to 100 weeks.
  Costs of nicotine replacement therapy will be captured using a single item added to the Cancer Patient Tobacco Use Questionnaire (item 15a)
Time between initial cancer diagnosis and administration of the DBT-ST intervention | Measured from the date of initial cancer diagnosis until week 1 of the patient's participation in the intervention, assessed up to 100 weeks.
  The impact on smoking cessation or reduction of the length of time between initial cancer diagnosis and administration of the DBT-ST intervention will be measured using the initial diagnosis date of any cancer per the patient's electronic health record and the Cancer Patient Tobacco Use Questionnaire
Group Size | Measured beginning 1 month after the date of week 8 of the final patient group participating in the intervention, assessed up to 6 months.
  The impact of group size on outcomes will be measured using the number of persons in each group, provided group size varies

CONTACTS AND LOCATIONS:
Overall Officials: Marcia McCall, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (2):
- United States (2):
  - Atrium Health Levine Cancer, Charlotte, North Carolina
  - Atrium Health Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: No